CLINICAL TRIAL: NCT02928900
Title: Simulated Patient Encounters to Promote Early Detection and Engagement in HIV Care for Adolescents
Brief Title: Patient Actor Training to Improve HIV Services for Adolescents in Kenya
Acronym: SPEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Nairobi (Other)
Responsible Party: Principal Investigator, Pamela Kohler, Assistant Professor, Global Health and Nursing, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002035
Record Dates: First submitted 2016-09-26; First posted 2016-10-10 (Estimated); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: HIV/AIDS
Keywords: Adolescents; Clinical training; HIV care and treatment; Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster RCT
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention period (Experimental): In this stepped-wedge trial design, the experimental arm refers to the time period when the study sites receive the clinician training intervention. The intervention is a clinician training using standardized patient actors to improve communication and empathy skills of health care providers who serve HIV-positive adolescents and youth.
  Interventions: Behavioral: Clinician training intervention
- Control period (No Intervention): In this stepped-wedge trial design, the no intervention arm refers to the time period before the study sites receive the clinician training intervention, during which standard of care is provided.

INTERVENTIONS:
Behavioral: Clinician training intervention — This intervention is a clinician training using SP actors to improve communication and empathy skills of HIV care providers who serve HIV-positive adolescents and youth in Kenya.
  Arms: Intervention period

SUMMARY:
The goal of this study is to develop and evaluate a clinical training intervention utilizing standardized patient actors to improve communication and interpersonal skills of health care workers who serve HIV-infected adolescents and youth in Kenya, resulting in increased engagement in HIV care. The effect of the intervention on retention in care will be evaluated in a stepped-wedge randomized controlled trial at 24 HIV care and treatment facilities.

DETAILED DESCRIPTION:
Adolescents and youth have the highest HIV incidence rates compared to any other age strata. Inadequate provision of accessible and acceptable HIV testing, counseling, and treatment services has been cited as a barrier to uptake of and retention in HIV care in this population.

The "SPEED" study aims to develop and evaluate a clinical training intervention utilizing Standardized Patient (SP) actors to improve communication and interpersonal skills of health care workers (HCWs) who work with adolescents and youth (ages 10-24), resulting in increased engagement in HIV care in Kenya. This intervention includes a series of role plays between HCW participants and professional Kenyan actors, followed by feedback and debriefing sessions. The hypothesis is that SP encounters will increase HCW confidence and capacity to facilitate HIV status disclosure and provide supportive interactions with HIV-infected youth, which will in turn increase uptake and improve retention in HIV services among adolescents and youth.

The pilot phase (Aim 1) will consist of developing patient case scripts specific to adolescent HIV-related care and counseling needs and establishing HCW competency scores. To evaluate the intervention, a cluster randomized controlled stepped-wedge trial will be conducted in 24 HIV care and treatment facilities to assess the impact of SP encounters on the proportion of adolescents and youth patients retained in care at HIV treatment facilities in Kenya (Aim 2). Finally, the cost effectiveness and cost utility of the SP intervention will be determined (Aim 3). The estimated study duration is five years.

The primary outcomes from Aim 1 are final scripts and pass/fail scores for use in SP encounters. The primary outcome for the randomized controlled trial (RCT) (Aim 2) is retention in care among HIV-positive adolescents and youth, based on electronic medical records data. Secondary outcomes will include satisfaction (patients and HCWs), HCW competency in youth- friendly counseling, antiretroviral therapy adherence, and viral suppression. For the cost effectiveness and cost utility analyses (Aim 3), the cost per additional HIV-infected adolescent/youth retained in care and the cost per additional life year saved and disability-adjusted life averted will be estimated.

ELIGIBILITY:
Inclusion Criteria: Listed by population

Facilities:

* HIV care and treatment facilities in Kenya with ≥40 adolescents currently in HIV care
* EMR data systems
* No concurrent adolescent interventions

Adolescent patient records:

* Records of adolescents and youth ages 10-24
* Enrollment in HIV care and treatment at one of the study facilities

Adolescent satisfaction surveys:

* Patients ages 10-24 seeking counseling or treatment services at trial site who are HIV-infected
* Willing and able to provide informed consent or assent based on age and presence of a caregiver.
* Reside in Kenya

Health care workers:

* >18 years of age
* Employed at trial site in clinical care for at least three months and/or have a 1 year contract (i.e. not temporary staff)
* Provide clinical services to adolescents
* Reside in Kenya

Exclusion Criteria:

Facilities:

* If inclusion criteria are not met
* If anything would prevent the complete conduct of the training intervention at that site and/or the collection of outcome measures

Adolescents and health care worker surveys:

• If an individual has conditions that would place them at increased risk or preclude the individual's full compliance with or completion of the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Kohler, PhD, MPH, RN, Principal Investigator — University of Washington; Dalton Wamalwa, MMed, MPH, Study Director — University of Nairobi
Locations (6):
- Kenya (6):
  - HIV care facility 6, Homa Bay
  - HIV care facility 3, Kiambu
  - HIV care facility 4, Kiambu
  - HIV care facility 5, Kisumu
  - HIV care facility 1, Nairobi
  - HIV care facility 2, Nairobi

IPD SHARING:
Plan to Share IPD: Yes
The study investigators are prepared to share data with other researchers in accordance with NIH policies and other local regulations.

REFERENCES:
- [Derived] Kohler PK, Mugo C, Wilson KS, Moraa H, Onyango A, Tapia K, Pike K, Mburu C, Nduati M, Guthrie B, Richardson BA, Owens T, Bukusi D, Inwani I, John-Stewart G, Wamalwa D. Simulated patient training to improve youth engagement in HIV care in Kenya: A stepped wedge cluster randomized controlled trial. PLOS Glob Public Health. 2023 Apr 19;3(4):e0001765. doi: 10.1371/journal.pgph.0001765. eCollection 2023. PMID 37074998
- [Derived] Wilson K, Onyango A, Mugo C, Guthrie B, Slyker J, Richardson B, John-Stewart G, Inwani I, Bukusi D, Wamalwa D, Kohler P. Kenyan HIV Clinics With Youth-Friendly Services and Trained Providers Have a Higher Prevalence of Viral Suppression Among Adolescents and Young Adults: Results From an Observational Study. J Assoc Nurses AIDS Care. 2022 Jan-Feb 01;33(1):45-53. doi: 10.1097/JNC.0000000000000302. PMID 34939987
- [Derived] Wilson KS, Mugo C, Bukusi D, Inwani I, Wagner AD, Moraa H, Owens T, Babigumira JB, Richardson BA, John-Stewart GC, Slyker JA, Wamalwa DC, Kohler PK. Simulated patient encounters to improve adolescent retention in HIV care in Kenya: study protocol of a stepped-wedge randomized controlled trial. Trials. 2017 Dec 28;18(1):619. doi: 10.1186/s13063-017-2266-z. PMID 29282109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stepped wedge design: 24 facilities randomized to when they received the training intervention. Once trained, all sites were considered intervention exposed for the duration of the study.
  De-identified adolescent medical records were analyzed for the primary outcome
Units Other Than Participants: HIV Clinics
Groups:
- Standardized Patient Training: Once assigned to the intervention, clinics received standardized patient actor training to improve quality of adolescent HIV care
- Control: Time period before exposure to training
Period: Baseline
Arm/Group | Standardized Patient Training | Control
Started (All 24 sites started as control sites. Sites were randomized to training in groups of 6 clinics every 9 months.) | NA; 0 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 24 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Completed | NA; 0 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 24 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Not Completed | NA; 0 HIV Clinics | NA; 0 HIV Clinics
Period: Wave 1
Arm/Group | Standardized Patient Training | Control
Started | NA; 6 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 18 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Completed | NA; 6 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 18 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Not Completed | NA; 0 HIV Clinics | NA; 0 HIV Clinics
Period: Wave 2
Arm/Group | Standardized Patient Training | Control
Started | NA; 12 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 12 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Completed | NA; 12 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 12 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Not Completed | NA; 0 HIV Clinics | NA; 0 HIV Clinics
Period: Wave 3
Arm/Group | Standardized Patient Training | Control
Started | NA; 18 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 6 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Completed | NA; 18 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 6 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Not Completed | NA; 0 HIV Clinics | NA; 0 HIV Clinics
Period: Wave 4
Arm/Group | Standardized Patient Training | Control
Started | NA; 24 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 0 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Completed | NA; 24 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records) | NA; 0 HIV Clinics (Arms were assigned based on clinic units. Outcomes assessed via de-identified patient records)
Not Completed | NA; 0 HIV Clinics | NA; 0 HIV Clinics

BASELINE CHARACTERISTICS:
Population: Clinics were assigned to the training intervention. Medical records were evaluated to assess study outcomes
Units Other Than Participants: Medical records
Groups:
- SP Training Intervention: HIV clinics were randomized to when they received the training intervention. The intervention consisted of a 2-day training for health providers at participating clinics. Once trained, all sites were considered intervention exposed for the duration of the study.
- No Training Intervention: Clinics prior to receiving training
- Total: Total of all reporting groups
Arm/Group | SP Training Intervention | No Training Intervention | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Medical records) | 2123 | 2472 | 4595
Age, Customized [Count of Units; unit: Medical records]
  10-14 | 220 | 278 | 498
  15-19 | 474 | 639 | 1113
  20-24 | 1429 | 1555 | 2984
Sex/Gender, Customized [Number; unit: Medical records]
  Female | 1761 | 2021 | 3782
  Male | 362 | 450 | 812
  Missing | 0 | 1 | 1
Race (NIH/OMB) [Count of Units; unit: Medical records]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2123 | 2472 | 4595
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Medical records]
  Kenya | 2123 | 2472 | 4595

OUTCOME MEASURES:

1. Primary Outcome: Retention in HIV Care
Description: The primary outcome is change in retention in HIV care between the intervention and control periods, where retention is defined as return for first follow-up visit within 3 months among newly enrolled adolescent clients OR follow-up visit after 're-engagement visit' (after lost-to-follow-up for >90 days since last visit, with no record of death or transfer).
Time Frame: Up to four years after baseline
Population: Medical record review. Final analysis accounts for clustering by facility, time (stepped wedge design), and newly enrolled in care status.
Measure: Count of Participants; unit: Participants
Groups:
- Adolescent Records - Intervention Exposed: Records from adolescents whose first eligible visit occurred at a facility that had already received the training intervention
- Adolescent Records - Unexposed: Records from adolescents whose first eligible visit occurred at a facility before the facility received the training intervention
Arm/Group | Adolescent Records - Intervention Exposed | Adolescent Records - Unexposed
Number analyzed (Participants) | 2123 | 2472
Participants | 1570 | 1855

2. Secondary Outcome: Proportion of HCWs With Pass/Fail Scores
Description: The proportion of HCW participants who achieved competency upon completion of the training.
Time Frame: Up to one month after last day of training
Reporting Status: Not Posted

3. Secondary Outcome: Numeric Scores From SP Actors
Description: All SP actors will complete a check-list to provide non-technical feedback to each HCW participant. Scores will be used to compute the overall pass/fail score at completion of the training.
Time Frame: Up to one week after last day of training
Reporting Status: Not Posted

4. Secondary Outcome: Health Care Worker Competency
Description: This outcome is measured as change in mean competency score between intervention and control periods using a structured survey.
Time Frame: Baseline and every nine months for up to four years
Reporting Status: Not Posted

5. Secondary Outcome: Health Care Workers' Satisfaction With Skills
Description: This outcome is measured as change in mean satisfaction scores between intervention (post-training) and control periods (pre-training), using a structured survey. These surveys will be conducted at baseline, and every nine months at the end of the training in each wave. Exit interviews among trained participants will be conducted about one year after each training wave for up to four waves to complement the quantitative results.
Time Frame: Baseline and every nine months for up to four years
Reporting Status: Not Posted

6. Secondary Outcome: Adolescent Patients' Satisfaction With Care
Description: This outcome is defined as mean change in satisfaction score between intervention and control periods, using a structured survey.
Time Frame: Baseline and every nine months for up to four years
Reporting Status: Not Posted

7. Secondary Outcome: Retention in HIV Care (Secondary)
Description: A secondary measure of retention in HIV care is return for any follow-up visit within 3 months (90 days) among currently enrolled HIV-positive adolescent patients
Time Frame: Baseline and every nine months for up to four years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Antiretroviral (ART) Adherence in HIV-positive Adolescents
Description: This measure is defined as change in the proportion of visits with ART refills within 1 week of scheduled visit between intervention and control periods using available electronic medical record (EMR) data.
Time Frame: Baseline and every nine months for up to four years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Viral Load in HIV-positive Adolescents
Description: This measure is defined as change in viral load between intervention and control periods using available EMR data.
Time Frame: Baseline and every nine months for up to four years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Linkage to Adolescent Friendly Services in HIV-positive Adolescents
Description: This measure is defined as change in the proportion of visits with referrals to affiliated services (e.g. family planning) between intervention and control periods using available EMR data.
Time Frame: Baseline and every nine months for up to four years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: AIDS Defining Illness in HIV-positive Adolescents
Description: This measure is defined as change in the proportion of visits with any AIDS defining illness between intervention and control periods using available EMR data.
Time Frame: Baseline and every nine months for up to four years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Mortality in HIV-positive Adolescents
Description: This measure is defined as change in the proportion of deaths between intervention and control periods using available EMR data.
Time Frame: Baseline and every nine months for up to four years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 years following the first intervention training.
Description: De-identified medical records are reported as the study population as they provided outcome data, however mortality data are largely missing in electronic records and the study was determined to be minimal risk (a health worker training program), thus we monitored for social harms related to counseling procedures and not post-training mortality among clients.
Groups:
- SP Training Intervention: In this stepped-wedge trial design, the experimental arm refers to the time period after study site clinicians receive the patient actor training intervention. All study sites eventually received the training intervention. Adolescents in the intervention arm presented for care after their site received training.
- No Training Intervention: In this stepped-wedge design, adolescents in the control arm presented for care before their site received training.
Arm/Group | SP Training Intervention | No Training Intervention
All-Cause Mortality (participants affected / at risk) | 0/2123 | 0/2472
Serious Adverse Events (participants affected / at risk) | 0/2123 | 0/2472
Other Adverse Events (participants affected / at risk) | 0/2123 | 0/2472

LIMITATIONS AND CAVEATS:
Data collection was suspended after Wave 4 training in March 2020 due to the COVID-19 pandemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02928900/Prot_SAP_000.pdf